CLINICAL TRIAL: NCT06894108
Title: The Effectiveness of a Proprietary of a Botanical Extract on Sleep Quality as Compared to a Melatonin Control: A Randomized, Double-Blinded, Controlled Clinical Trial
Brief Title: The Effectiveness of a Proprietary of a Botanical Extract on Sleep Quality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nutraceuticals Research Institute (Other)
Responsible Party: Principal Investigator, Jessie Hawkins, Primary Investigator, Nutraceuticals Research Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 24-05-500
Record Dates: First submitted 2025-03-19; First posted 2025-03-25 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Sleep
MeSH Terms: interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Botanical Blend (Experimental)
  Interventions: Dietary Supplement: Proprietary Blend of Botanical Extracts
- Comparison (Active Comparator)
  Interventions: Dietary Supplement: Melatonin

INTERVENTIONS:
Dietary Supplement: Proprietary Blend of Botanical Extracts — Participants consumed 2.4ml of the supplement each night before bed.
  Arms: Botanical Blend
Dietary Supplement: Melatonin — Participants consumed 1mg melatonin each night before bed.
  Arms: Comparison

SUMMARY:
The purpose of this study is to evaluate the efficacy and superiority of a botanical based sleep product on sleep quality as compared to melatonin, among healthy female participants.

ELIGIBILITY:
Inclusion Criteria:

Provision of signed and dated informed consent form Stated willingness and demonstrated ability to comply with all study procedures, as well as availability for the duration of the study Self reported poor sleep quality Biological sex of woman; gender identification of female Aged 35 to 55, inclusive Good general health as evidenced by medical history and screening For females of reproductive potential: use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation and for an additional month after the end of the study Has an apple watch or similar device Agreement to adhere to Lifestyle Considerations throughout study duration

Exclusion Criteria:

Pregnancy, trying to conceive, or breastfeeding Currently smokes or vapes (i.e., tobacco, flavored items, marijuana, etc.) or has in the past year Has received medical diagnosis or treatment for any sleep disorder in the past year Has ever received a medical diagnosis of sleep apnea or narcolepsy Works a night shift, is "on-call" or performs any job requiring or potentially requiring work related responsibilities after 8pm Consumes > 8 alcoholic beverages in an average week Is a primary caretaker for a child younger than 18 months of age Consumes any sleep aid, medication, diet, or supplement intended to improve sleep in any way Known allergic reactions to any components of the intervention Positive COVID-19 test within 30 days of the study period Recent dramatic weight changes (10% change in body weight in the last 6 months) Introducing a new investigational drug or other intervention within 60 days before the start of the study

Ages: 35 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Individuals who identify as female quality to participate.
Enrollment: 89 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
NRI Sleep Scale | From baseline to the end of the 28 day intervention.
  The NRI Sleep Scale is a validated measure of sleep health. It has 6 domains, each measured on a Likert scale, with higher scores indicating greater sleep disturbances.

SECONDARY OUTCOMES:
Wearable Technology | From baseline to the end of the 28 day intervention.
  Sleep data sourced from the participant's Apple Watch (time in bed, time spent per phase (awake, REM, core, and deep).
NRI Energy Scale | From baseline to the end of the 28 day intervention.
  Description: The NRI Energy Scale is a validated measure of fatigue. It has 7 domains, each measured on a Likert scale, with higher scores indicating greater fatigue.

CONTACTS AND LOCATIONS:
Locations (1):
- Nutraceuticals Research Institute, Huntsville, Alabama, United States

IPD SHARING:
Plan to Share IPD: No